CLINICAL TRIAL: NCT02629276
Title: Somatosensory Profiles in Patients With Non Specific Neck Arm Pain With and Without Positive Neurodynamic Tests
Brief Title: Somatosensory Phenotype of Patients Suffering From Unspecific Neck and Arm Pain
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2014-12
Record Dates: First submitted 2015-12-07; First posted 2015-12-14 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Neck Pain
Keywords: neck pain; arm pain; neurodynamic tests; quantitative sensory testing; somatosensory profile
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: neurodynamic testing

SUMMARY:
The aim of this study was to evaluate potential differences in somatosensory function in patients with unilateral NSNAP with and without positive ND compared to healthy controls. Furthermore, we determined whether there are any differences between groups in symptom severity, functional deficits, psychological parameters, quality of life and sleep.

DETAILED DESCRIPTION:
Neck pain is a common musculoskeletal problem, with up to 30-50 % of adults experiencing neck pain in any given year. Neck pain in combination with arm pain is more common than neck pain alone and is associated with higher Ievels of self-reported disability and psychological impairment. In most cases, no pathophysiological correlate can be found in various investigations including magnetic resonance imaging of the cervical spine and tests for nerve conductivity (bedside neurological examination and standard electro diagnostic tests). In such cases, the neck-arm pain is labelled as non-specific. Although clinical examinations that evaluate the conductivity of the nervous system are normal in non-specific neck-arm pain (NSNAP), neurodynamic tests (ND) have been identified as positive in a subgroup of patients. ND are clinical tools designed to elongate the nerve bed, therefore increasing the mechanical loading of neural tissues. As such, ND provide information about alterations of neural tissue mechanosensitivity, i.e. the presence of heightened nerve mechanosensitivity. It is assumed that increased neural mechanosensitivity reflects gain of function, presumably mediated by small nociceptive fibres intraneurally or within the epineurium (nervi nervorum). However, it remains unclear whether the subgroup of patients with NSNAP and positive ND have indeed increased gain of function of this small fibre population compared to those patients with normal ND.

Quantitative sensory testing (QST) is a commonly used tool to determine the function of different subsets of small (C, Ad-fibres) and large nerve fibres (Ad-fibres). Using QST, a recent study has identified a loss of small fibre function in patients with unilateral NSNAP and positive ND as apparent by reduced warm detection thresholds compared to the non-affected side. However, this difference was small and potentially not clinically rele-vant and the relatively small sample size of n=8 does not allow generalization of the results. In the same study, patients with NSNAP were also characterized by a gain of function, i.e. cold hypersensitivity. Similarly, widespread thermal and pressure hypersensitivity have been documented in patients with nonspecific arm pain (with or without neck pain). None of these studies has however investigated a potential difference between patients with NSNAP with positive versus negative ND, leaving it unclear whether the QST findings can indeed be attributed to a positive ND.

A recent study compared patients with NSNAP and neuropathic features using ND testing and a self report neuropathic pain screening tool and patients with NSNAP and no neuropathic features. Interestingly, the first group showed heightened nerve mechanosensitivity apparent by an earlier onset of symptoms during ND testing. This raises the question whether patients with NSNAP and positive ND have indeed a dysfunction of their nervous system that differentiates them from patients with normal ND.

ELIGIBILITY:
Inclusion Criteria:

- unilateral non specific neck-arm pain

Exclusion Criteria:

* specific neck-arm pain (e.g., cervical radiculopathies, myelopathies)
* underlying diseases (e.g, central neurological condition, metabolic disease)
* upper limb or spinal surgery or significant trauma in the preceding two years
* manifest psychiatric or mental diseases
* insufficient German language skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (woman and men) with unilateral non specific neck-arm pain are recruited from the Centre of Pain Medicine outpatient departments of the Swiss Paraplegic Centre in Nottwil. A standard bedside neurological examination (light touch, muscle strength and reflexes) and standard electro-diagnostic tests (distal ulnar and median sensory and motor latencies and amplitudes, F-waves) are performed to exclude patients with a specific neurological cause for their symptoms (e.g., cervical radiculopathies, myelopathies)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
mechanosensitivity of neural tissue in neurodynamic testing | at enrolment

SECONDARY OUTCOMES:
sensation thresholds for cold and warm temperatures in quantitative sensory testing | at enrolment
pain thresholds for cold and warm temperatures in quantitative sensory testing | at enrolment
vibration sensation threshold in quantitative sensory testing | at enrolment
disability due to neck pain | at enrolment
  neck disability index questionnaire
presence of neuropathic pain | at enrolment
  neuropathic pain symptom inventory questionnaire
presence of anxiety | at enrolment
  hospital anxiety and depression scale questionnaire
presence of depression | at enrolment
  hospital anxiety and depression scale questionnaire
insomnia severity | at enrolment
  insomnia severity index questionnaire
sleep quality | at enrolment
  visual analogue scale
presence of pain catastrophizing | at enrolment
  pain catastrophizing scale questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gunther Landmann, Study Director — Swiss Paraplegic Centre
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No